CLINICAL TRIAL: NCT06763523
Title: Arthroereisis With Corrective Osteotomy Versus Arthroereisis Alone in Management of Symptomatic Flexible Pes Planovalgus in Adolescents
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ahmed Mohy Eldien Abdelrahman, Specialist, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Soh-24-12---1MD
Record Dates: First submitted 2024-12-23; First posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Pes Plano Valgus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group B (Active Comparator): arthroereisis without corrective osteotomies
  Interventions: Procedure: arthroereisis of the subtalar joint
- Group A (Active Comparator): arthroereisis with corrective osteotomies
  Interventions: Procedure: arthroereisis of the subtalar joint

INTERVENTIONS:
Procedure: arthroereisis of the subtalar joint — arthroereisis alone versus arthroereisis combined with corrective osteotomies

SUMMARY:
Arthroereisis ,corrective osteotomies, flexible pes planovalgus, adolescents

ELIGIBILITY:
Inclusion Criteria:

* cases complaining of flexible pes planovalgus non responsive for conservative treatment and cases with generalized ligamentous laxity

Exclusion Criteria:

* neurological disorders and rigid peaplanovalgus

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2025-01-19 (Estimated); Primary Completion 2025-01-20 (Estimated); Study Completion 2026-01-20 (Estimated)

PRIMARY OUTCOMES:
AOFAS score | 2 years from the start of the study
  American Orthopaedic Foot & Ankle Society

SECONDARY OUTCOMES:
VAS score | 2 years from the start of the study
  visual analog score

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided